CLINICAL TRIAL: NCT00063596
Title: Vitamin A Therapy in Preterm Infants: Vaccine Response
Brief Title: Vitamin A Supplementation in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01HD037263 (NIH)
Record Dates: First submitted 2003-07-01; First posted 2003-07-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-11

CONDITIONS: Infant, Premature
Keywords: Vitamin A; Hepatitis B vaccine; Immune responses; T-cell subsets; Chronic lung disease; Cytokines, intracytoplasmic; Antibodies, hepatitis B and tetanus toxoid
MeSH Terms: conditions — Premature Birth; Hepatitis B; Tetanus

INTERVENTIONS:
Drug: Vitamin A supplementation

SUMMARY:
Extremely low birth weight infants have decreased blood levels of Vitamin A. This Vitamin A deficiency may increase the risk of infections and chronic lung disease in these infants. This study will examine the effects of Vitamin A supplementation in premature babies born weighing less than 1500 grams (3.3 lbs).

DETAILED DESCRIPTION:
Vitamin A and its derivative retinoic acid (RA) have been recognized as important factors in potentiating the immune response and protecting against infection. In developing nations, Vitamin A deficiency is associated with infectious gastroenteritis and increased susceptibility to a number of infections, such as measles. RA is an important regulator of cell growth and differentiation and can augment IgM production from core blood mononuclear cells in response to a polyclonal B-cell activator. This augmentation in immunoglobulin secretion is mediated by the effects of RA on both T and B cells, in part through the production of certain cytokines (e.g., IL-6 and IL-10) important in the terminal differentiation of B-cells to plasma cells. In animal models, correction of Vitamin A deficiency improves immune response to vaccination.

Infants with extremely low birth weight have low plasma and tissue concentrations of Vitamin A. Vitamin A supplementation of pre-term infants reduces chronic lung disease and the risk of sepsis. Because the immune system of the pre-term infant is immature, the response of pre-term infants to Hepatitis B vaccine is diminished compared to full-term babies. This study will determine whether Vitamin A supplementation of pre-term infants will enhance the response of these infants to immunization with Hepatitis B vaccine. The study will also evaluate the effect of Vitamin A supplementation on survival, chronic lung disease, and infection rate.

Low birth weight pre-term infants will be randomized to receive either Vitamin A supplementation or placebo. The Vitamin A treatment group will receive 5,000 IU of Vitamin A (retinyl palmitate) by intramuscular injection 3 times weekly for 28 days starting on postnatal day 2. To avoid pain and discomfort, the placebo group will receive a sham procedure rather than a placebo saline injection. The staff of the neonatal intensive care unit will retain the responsibility for decisions regarding the use of other therapies, such as parental fluids, mechanical ventilation, glucocorticoids, hyperalimentation, and blood replacement. All infants will be assessed for potential Vitamin A toxicity. While in the neonatal intensive care unit, infants will have blood tests at Days 0, 14, 30, and 60. After discharge from the neonatal intensive care unit, patients return for clinic assessment and blood samples at Months 4, 6, and 9. Infants will be given Hepatitis B vaccine at 2, 4, and 6 months chronological age. Primary outcome measures will include Hepatitis B antibody levels, chronic lung disease, rate of infection while in the neonatal intensive care unit, and the incidence and severity of infections during the first 9 months of life.

ELIGIBILITY:
Inclusion Criteria

* Born at less than 32 weeks gestation
* Weigh less than 1500 g (3.3 lbs) and more than 500 g (1.1 lbs)

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220
Dates: Start 2000-01; Study Completion 2004-05

PRIMARY OUTCOMES:
Response to Hepatitis B vaccine

SECONDARY OUTCOMES:
Chronic lung disease
Length of hospital stay
Respiratory and GI infections to 9 months of age
T-cell cytokine production and development
T-cell subset development

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ballow, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Women's and Children's Hospital of Buffalo, Buffalo, New York, United States